CLINICAL TRIAL: NCT01557621
Title: Center for Research in Implementation Science and Prevention (CRISP): Project 1: Comparative Effectiveness Trial of Two Reminder/Recall Methods to Increase Immunization Rates in Young Children
Brief Title: Comparative Effectiveness Trial of Two Reminder/Recall Methods to Increase Immunization Rates in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 11-1480; P01HS021138 (AHRQ)
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Immunization Rates
Keywords: Immunization reminder/recall; Reminder/Recall systems; Population based Recall; Practice based Recall

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Collaborative Population-Based Recall-Phone/Mail Group (Experimental): Collaborative Pop-Based R/R: Phone/Mail Group Private providers, local public health departments, and the state immunization registry (CIIS) collaborate to send notices to families whose children appear in need of an immunization.
  Interventions: Behavioral: Collaborative Pop-Based R/R: Phone/Mail Group
- Collaborative Population-Based Recall-Mail Only Group (Experimental): Collaborative Pop-Based R/R: Mail-Only Group Private providers, local public health departments, and the state immunization registry (CIIS) collaborate to send notices to families whose children appear in need of an immunization.
  Interventions: Behavioral: Collaborative Pop-Based R/R: Mail-Only Group
- Practice-based Recall (Active Comparator): Practice-based Recall
  Interventions: Behavioral: Practice-based Recall

INTERVENTIONS:
Behavioral: Collaborative Pop-Based R/R: Phone/Mail Group — Within each county, half of patients will be randomized to a phone/mail group (2 auto-dialer calls and 2 postcards) and the other half of patients will be put in a mail-only group (4 mailings). The following collaborative approaches will be utilized: patient addresses and phone numbers will be updated prior to recall for electronic Flat File Format practices; all notices to parents (auto-dialer calls and mailings) will appear to come both from the local public health department and providers who choose to have their name listed; all bad addresses and phone numbers will be updated by calling the last provider of care. Up to 4 notices will be sent to parents of children who are still not up to date for recommended immunizations.
  Arms: Collaborative Population-Based Recall-Phone/Mail Group
Behavioral: Collaborative Pop-Based R/R: Mail-Only Group — Parents will receive up to four mailings if their child appears in need of immunizations according to CIIS. The Collaborative method is the same as in the auto-dialer/mail group; however patients in this group will not receive telephone calls.
  Arms: Collaborative Population-Based Recall-Mail Only Group
Behavioral: Practice-based Recall — All practices will receive training on how to conduct practice-based recall using CIIS and educational materials to use within their practices to promote compliance with the infant vaccination schedule. Individual practices will make their own decisions about the extent to which they follow the recommendations and implement recall within their practice. Although the study team will not provide them with any additional interventions, we will track any other interventions they independently do (websites, newsletters, telephone) in order to assess the effect of these additional interventions.
  Arms: Practice-based Recall

SUMMARY:
The purpose of this study is to determine if a collaborative centralized population-based reminder/recall intervention is more effective than a traditional practice-based reminder/recall intervention at increasing immunizations among young children.

DETAILED DESCRIPTION:
The study proposed is of immense importance in directing future methodology for bringing children who have not received needed immunizations up to date. The proposed study builds on the success of a previous trial and incorporates data from providers and patients to further improve the intervention. In this study the investigators aim to increase the effectiveness, cost effectiveness, and acceptability to practices and families of population-based R/R by introducing a strong private-public collaboration and maximizing health information technologies that allow practices to interface with Colorado's Immunization Services System (CIIS). Two real-world approaches will be compared: one approach will provide primary care practices the tools to conduct recall and educational interventions. In the other approach, population-based centralized recall by the state immunization registry will be conducted in collaboration with practices. Determining which of these methods is most effective in reaching the most children and comparing the cost of each will provide data critical in guiding future national efforts to assure that children entering school are fully vaccinated. Because the trial will be conducted at the level of both urban and rural counties throughout the state and will include all types of providers, the investigators expect our findings to be nationally generalizable.

ELIGIBILITY:
Inclusion Criteria:

* 19-35 months at time of recall
* has an address in a specified study county listed in the state immunization registry
* child is in need of at least one immunization at time of study

Exclusion Criteria:

* Opted out of the Colorado Immunization Information System (CIIS)
* child is up-to-date on all immunizations

Ages: 19 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68000 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
1) Change in up-to-date rates for 19- to 35-month-olds (who needed an immunization at baseline) in collaborative population-based counties compared to practice-based intervention counties | every 6 months for 2 years
  The definition of up-to-date is based on the national Advisory Committee on Immunization Practices(ACIP)recommended series of antigens (4:3:1:3:3:1:3) to be received by the age of 19-20 months. Three different cohorts of children aged 19-35 months will be assessed across the 3 year study period. Outcomes from each cohort will be assessed 6 months post-intervention.
2) Change in percent of children (who needed an immunization at baseline) who received any additional vaccines in each type of intervention county. | every 6 months for two years
  Number (percent) of children who received ANY vaccination within the 6 month intervention period.

SECONDARY OUTCOMES:
Cost Analysis of Collaborative Population-based Recall versus Practice-based Recall | 2 years
  Number (percent) of identified children that became up-to-date for recommended immunizations.
  Number (percent) of shots delivered to children needing immunizations. Number (percent) or providers (sites) that conducted practice-based reminder recall.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kempe, MD, MPH, Principal Investigator — University of Colorado Denver, The Children's Hospital of Colorado
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - Colorado Immunization Information System, Denver, Colorado

REFERENCES:
- [Derived] Kempe A, Saville AW, Dickinson LM, Beaty B, Eisert S, Gurfinkel D, Brewer S, Shull H, Herrero D, Herlihy R. Collaborative centralized reminder/recall notification to increase immunization rates among young children: a comparative effectiveness trial. JAMA Pediatr. 2015 Apr;169(4):365-73. doi: 10.1001/jamapediatrics.2014.3670. PMID 25706340